CLINICAL TRIAL: NCT00578461
Title: T-Regulatory Cell Kinetics Post Transplant For Patients Undergoing Matched Sibling Stem Cell Transplantation
Brief Title: T-Regulatory Cell Kinetics, Stem Cell Transplantation, REGKINE
Acronym: REGKINE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Robert Krance, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-19164 REGKINE; NCT00653289 (obsolete NCT alias)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-03

CONDITIONS: Leukemia; Cancer; Lymphoma; Lymphoma, Hodgkin; Lymphoma, Non-Hodgkin
Keywords: Stem Cell Transplant; myeloproliferative disease; myelodsyplastic disease; Leukemia; Cancer; Lymphoma; Lymphoma, Hodgkin; Lymphoma, non-Hodgkin
MeSH Terms: conditions — Leukemia; Neoplasms; Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Myeloproliferative Disorders | interventions — Cytarabine; Mesna; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell Transplant (Experimental): patient's will be recieving a stem cell transplant on study Conditioning includes: Ara C, Cyclophosphamide, MESNA, TBI-Total Body Irradiation
  Interventions: Drug: Ara C; Drug: Mesna; Drug: Cyclophosphamide; Radiation: TBI-Total Body Irradiation

INTERVENTIONS:
Drug: Ara C — 3000 mg/m^2 - pts will recieve via IV every 12 hours for 6 doses starting at 20:00 hours on day -8
  Other Names: Cytarabine; Cytosar-U
Drug: Mesna — 45 mg/kg; divided into 5 doses-will be administered 15 minutes prior to Cyclophosphamide and 3, 6, 9, and 12 hours after each dose of Cyclophosphamide
  Other Names: Mesnex
Drug: Cyclophosphamide — 45 mg/kg; IV once daily on day -7 and day -6 starting at 1400 hours
  Other Names: Cytoxan
Radiation: TBI-Total Body Irradiation — Total dose 12 Gy, will be delivered in 8 fractions of 150 cGy, each, two fractions per day beginning day -4

SUMMARY:
Patients are being asked to participate in this study because they have a cancer in their blood (such as leukemia or lymphoma) or myelodysplastic/myeloproliferative (pre-leukemia). We suggest a treatment that might help them live longer without disease than other treatment plans would. This treatment is known as a stem cell transplant. We believe this may help the patient as it allows us to give much stronger doses of drugs and radiation to kill the diseased cells than we could give without the transplant. We also think that the healthy cells may help fight any diseased cells left after the transplant.

Stem Cells are special "mother" cells that are found in the bone marrow (the spongy tissue inside bones), although some are also found in the bloodstream (peripheral blood). As they grow, they become either white blood cells which fight infection, red blood cells which carry oxygen and remove waste products from the organs and tissues or platelets, which enable the blood to clot. For the transplant to take place, we will collect these stem cells from a "donor" (a person who agrees to donate these cells) and give them to the patient. The patient has a type of blood cell cancer or other blood problem that is very hard to cure with standard treatments and they will receive a stem cell transplant (SCT). If they have a brother or sister that is a perfect match and agrees to donate, the stem cells will come from him/her. Before the transplant, two very strong drugs plus total body irradiation will be given to the patient (pre-conditioning). This treatment will kill most of the blood-forming cells in the bone marrow. We will then give the patient the healthy stem cells. Once these healthy stem cells are in the bloodstream they will move to the bone marrow (graft) and begin producing blood cells that will eventually mature into healthy red blood cells, white blood cells and platelets.

Also, we will ask permission to draw blood from the patient so that we can measure the number of certain blood cells called T regulatory cells. T regulatory cells are special immune cells that can control or regulate the body's immune response. We want to determine whether T regulatory cells are important participants in graft versus host disease (GVHD), infection and relapse. In GVHD, certain cells from the donated marrow or blood (the graft) attack the body of the transplant patient (the host). GVHD can affect many different parts of the body. The skin, eyes, stomach and intestines are affected most often. GVHD can range from mild to life-threatening. We do not know whether T regulatory cells can modify these conditions. We want to measure these T regulatory cells and learn if these cells do influence these conditions. If we learn that T regulatory cells do affect these conditions, then it may be possible to modify these cells for the benefit of transplant patients.

DETAILED DESCRIPTION:
Before the transplant we will test the patients blood for viruses which can cause problems after the transplant. These viruses include Hepatitis B, (which causes liver damage), cytomegalovirus, (which causes lung disease) and HIV (which causes AIDS). If the patient is positive for the AIDS virus, they will not be able to undertake the transplant.

The patient will be given 6 doses of chemotherapy with a drug called Ara C in high doses (every 12 hours) which will begin 8 days before their stem cell transplant. Then, another chemotherapy drug called cyclophosphamide will be given in high doses by vein for two days on the 7th and 6th days before their transplant. A drug called MESNA will be given with cyclophosphamide. MESNA is used to decrease the side effects caused by cyclophosphamide. Radiation treatment will be given to the entire body on each day for 4 days before the transplant. This will be done 2 times a day for 4 days. The chemotherapy and radiation treatment will last 8 days. The patient will receive extra radiation treatment if they have certain diseases (central nervous system (CNS) disease, testicular disease or other focal (localized) disease).

The day after the radiation treatment is completed; the patient will receive the healthy stem cells by vein. Once in the bloodstream, these stem cells will go to the bone marrow and should begin to grow

In prevention of GVHD, the patient will also receive medicine called FK506 as well as low dose methotrexate. The FK506 will be given intravenously (through the vein) initially starting 2 days before the transplant and later by mouth (when they are able to take oral medications). This drug will be given each day for several weeks. Four doses of low dose methotrexate will be given intravenously. The methotrexate will be given on the day after the transplant, 3, 6 and 11 days after the transplant. If the GVHD cannot be controlled with FK506, other medicines may need to be given. Your doctor will describe these medicines at that time.

After the patient has their stem cell transplant, we would like to collect some blood at different time points after the transplantation in order to study how regulatory T cells work and grow after a stem cell transplant.

To study how these cells are working in the system, blood samples will be taken each month for six months, at nine months, at one year, 2 years and 3 years following transplant. Approximately 6-8 teaspoons of blood will be collected each time. The total blood drawn for this study over three years should not exceed 1 and 3/4 cups. This amount is considered safe in adults. The amount of blood collected will be decreased in children and/or in patients where this amount of blood collection would not be appropriate. If the patient has a central line, the blood will be taken from it, so that extra needle sticks should not be needed. If the patient does not have a central line, they will need to have one placed. This will be a separate procedure for which the patient will sign a separate consent form. The patient will need to come to the clinic on the days of blood drawing and to be seen at Texas Children's Cancer Center.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with acute or chronic leukemia or advanced Hodgkin or non Hodgkin lymphoma or myelodysplastic/myeloproliferative disease who are unlikely to be cured by standard chemotherapy treatments. This includes patients who have relapsed after standard chemotherapy treatments and patients in first remission with unfavorable prognostic features.
* Patient must have a genotype HLA identical stem cell donor.

EXCLUSION CRITERIA:

* Patients with a life expectancy (less than or equal to 6 weeks) limited by disease other than leukemia.
* Patients with symptomatic cardiac failure unrelieved by medical therapy or evidence of significant cardiac dysfunction by echocardiogram (shortening fraction <20%).
* Patients with severe renal disease (i.e., creatinine greater than 3 times normal for age).
* Patients with pre-existing severe restrictive pulmonary disease (FVC less than 40% of predicted).
* Patients with severe hepatic disease (direct bilirubin greater than 3 mg/dl or AST greater than 500 IU/L).
* Patients with severe personality disorder or mental illness.
* Patients with severe infection that in the estimation of the principal investigator prohibits the use of ablative chemotherapy.
* Patients who are documented HIV positive.
* Patients with a Karnofsky performance score <60% or Lansky performance score <50%.

NOTE: Patients who would be excluded from treatment on this protocol strictly for laboratory or performance abnormalities can be included at the principal investigator's discretion after consultation with the members of the SCT Policy and Procedures Committee.

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2007-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krance, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Stem Cell Transplant: All patients will receive stem cell transplantation conditioning, GVHD prevention and stem cell infusion.
  Conditioning includes: Ara C, Cyclophosphamide, MESNA, TBI-Total Body Irradiation. Ara C: 3000 mg/m^2 - pts will receive via IV every 12 hours for 6 doses starting at 20:00 hours on day -8.Mesna: 45 mg/kg; divided into 5 doses-will be administered 15 minutes prior to Cyclophosphamide and 3, 6, 9, and 12 hours after each dose of Cyclophosphamide.
  Cyclophosphamide: 45 mg/kg; IV once daily on day -7 and day -6 starting at 1400 hours.TBI-Total Body Irradiation: Total dose 12 Gy, will be delivered in 8 fractions of 150 cGy, each, two fractions per day beginning day -4 to day -1. Stem cell Infusion is on day 0.
Period: Overall Study
Arm/Group | Stem Cell Transplant
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 26 patients were enrolled on the study and all of them received the conditioning treatment and the transplant.
Groups:
- Stem Cell Transplant: All patients will receive stem cell transplantation conditioning, GVHD prevention and stem cell infusion.
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (4.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Median Percentage of Treg Cells at 1 Year Post Transplant
Description: The investigative intent is to determine the changes in numbers and function of the regulatory cell population using the best methods to measure this cell population. The frequency of T cells will be summarized at baseline and each time point of follow-up.
Time Frame: 1 Year
Population: Only 20 of the 26 patients enrolled were included in this analysis as only 20 patients have Treg values at 1 year.
Measure: Median (Inter-Quartile Range); unit: percentage of total CD4+ cells
Groups:
- Stem Cell Transplant: All patients will be receiving a stem cell transplant on study. Conditioning includes: Ara C, Cyclophosphamide, MESNA, TBI-Total Body Irradiation.
Arm/Group | Stem Cell Transplant
Number analyzed (Participants) | 20
percentage of total CD4+ cells | 4.1 [3.1 to 6.4]

ADVERSE EVENTS:
Arm/Group | Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 15/26
Other Adverse Events (participants affected / at risk) | 16/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Transplant (N=26)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 2 (3)
Coagulation - Other: Severe coagulopathy (Vascular disorders) | 1 (1)
Fever (General disorders) | 1 (2) — Fever in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L
Death (General disorders) | 1 (1) — Death is not associated with CTCAE term - Multi-organ failure
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 2 (3)
Febrile neutropenia (Infections and infestations) | 1 (1) — Fever of unknown origin without clinically or microbiologically documented infection. ANC <1.0 x 10e9/L, fever >=38.5 degrees C.
Infection with Grade 3 or 4 neutrophils - Catheter-related (Infections and infestations) | 1 (2) — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Catheter-related
Infection with Grade 3 or 4 neutrophils - Vein (Infections and infestations) | 1 (1) — Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - Vein
Infection - Other: only clinical signs of infection (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Catheter-related (Infections and infestations) | 5 (6)
Infection with normal ANC or Grade 1 or 2 neutrophils - Nose (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 1 (1)
AST, SGOT (Metabolism and nutrition disorders) | 1 (1) — SGOT: serum glutamic oxaloacetic transaminase
Pain - Abdomen NOS (General disorders) | 1 (1)
Pain - Head/headache (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (4)
Portal vein flow (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Transplant (N=26)
PTT (Vascular disorders) | 2 (3) — PTT: Partial Thromboplastin Time
Diarrhea (Gastrointestinal disorders) | 4 (4)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (5)
Infection with normal ANC or Grade 1 or 2 neutrophils - Catheter-related (Infections and infestations) | 3 (3)
ALT, SGPT (Metabolism and nutrition disorders) | 2 (2) — SGPT: serum glutamic pyruvic transaminase
AST, SGOT (Metabolism and nutrition disorders) | 4 (6) — SGOT: serum glutamic oxaloacetic transaminase
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2)
GGT (Metabolism and nutrition disorders) | 2 (2) — GGT: gamma-Glutamyl transpeptidase
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes